CLINICAL TRIAL: NCT02100852
Title: A Multi-center Phase I/Ib Study Evaluating the Efficacy and Safety of TGR-1202, a Novel PI3K Delta Inhibitor, in Combination With Obinutuzumab and Chlorambucil in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: TGR-1202, a PI3K Delta Inhibitor, in Combination With Obinutuzumab and Chlorambucil in Patients With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGR-GA-106
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — umbralisib; obinutuzumab; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TGR-1202 + Obinutuzumab + Chlorambucil (Experimental): TGR-1202 is an oral daily dose with obinutuzumab at a fixed IV infusion and chlorambucil as an oral dose on specified days.
  Interventions: Drug: TGR-1202 + Obinutuzumab + Chlorambucil

INTERVENTIONS:
Drug: TGR-1202 + Obinutuzumab + Chlorambucil — TGR-1202: Oral dose Obinutuzumab: IV infusion Chlorambucil: Oral dose
  Other Names: Obinutuzumab: Gazyva; Chlorambucil: Leukeran

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of TGR-1202 in combination with obinutuzumab (Gazyva) and chlorambucil in patients with chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Chronic Lymphocytic Leukemia (CLL)
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2
* Ability to swallow oral medication

Exclusion Criteria:

* Known hepatitis B virus, hepatitis C virus or HIV infection
* Primary central nervous system lymphoma or known intracranial involvement
* Autologous hematologic stem cell transplant within 3 months of study entry or Allogeneic hematologic stem cell transplant within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose acceptable for participants | 28 days (1 cycle of therapy)
  To determine the incidence of adverse events, any potential abnormal laboratory results and any dose-limiting toxicities

SECONDARY OUTCOMES:
Overall Response Rate | Up to 1 year
  To assess the overall response rate (ORR) in patients with chronic lymphocytic leukemia treated with TGR-1202 in combination with obinutuzumab (Gazyva) and chlorambucil

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Memphis, Tennessee